CLINICAL TRIAL: NCT03400059
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter Study to Evaluate the Efficacy of Intranasal Kinetic Oscillation Stimulation in the Preventive Treatment of Chronic Migraine
Brief Title: Study to Evaluate the Efficacy of Intranasal Kinetic Oscillation Stimulation in the Preventive Treatment of Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chordate Medical (Industry)
Collaborators: Vinnova (Other Government); FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PM007
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Chronic Migraine
Keywords: Prophylaxis, Headache, Preventative Treatment
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental)
  Interventions: Device: Chordate System S211 in treatment mode
- Sham Treatment (Sham Comparator)
  Interventions: Device: Chordate System S211 in placebo mode

INTERVENTIONS:
Device: Chordate System S211 in treatment mode — Chordate System S211 in treatment mode
  Arms: Active Treatment
Device: Chordate System S211 in placebo mode — Chordate System S211 in placebo mode
  Arms: Sham Treatment

SUMMARY:
The efficacy of intranasal kinetic oscillation stimulation using the Chordate System S211 as a preventative treatment will be examined in patients diagnosed with chronic migraine. The medical device system will be applied in 6 treatments at weekly intervals. The study will examine the effects on monthly headache days with moderate to severe intensity.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multicenter clinical investigation of a medical device. The study consists of a 4-week screening period, a 6-week treatment period (2 weeks run-in and a 4-week observation window to assess the treatment effect), and a 4-week follow-up period.

The study primarily aims at evaluating the effect of intranasal kinetic oscillation stimulation using the Chordate System S211 as a preventative treatment on monthly headache days with moderate to severe intensity.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the informed consent form (ICF);
2. Male or female aged between 18 and 65 years (inclusive) at the time of providing informed consent;
3. Diagnosed as suffering from chronic migraine with or without aura (≥15 headache days per month for more than 3 months before screening including at least 8 migraine days) according to the IHS classification (International Classification of Headache Disorders [ICHD]-III beta);
4. Migraine onset before the age of 60 years;
5. Reported history of migraine for at least 1 year before screening;
6. Reported stable prophylactic migraine medication regimen, if any, during the 3 months prior to screening;
7. Able and willing to maintain current prophylactic migraine medication regimen (no change in type, frequency or dose) from screening to end of follow-up;
8. Women of childbearing potential must be willing to use highly effective contraceptive methods (failure rate <1% per year when used consistently and correctly) during the study.

Exclusion Criteria:

1. Unable to distinguish between migraine headaches and other headache types;
2. Treatment with Botox in the head/neck area within 4 months of the screening visit, or planned Botox treatment during the study;
3. Previous or ongoing treatment with an implanted stimulator or other implanted device in the head and/or neck;
4. Known pronounced anterior septal deviation, or other known relevant abnormality in the nasal cavity, including bacterial infection and wounds;
5. History of relevant sinus surgery, transsphenoidal surgery for pituitary or other lesions or cerebrospinal fluid (CSF) rhinorrhea;
6. Fitted with a pacemaker/defibrillator;
7. Previously treated with therapeutic x-ray intervention in the facial region (that could have influenced the nasal mucosa);
8. Ongoing upper respiratory infection or malignancy in the nasal cavity;
9. History of regular nose bleeding (epistaxis), or concomitant condition or medication that could cause excessive bleeding including treatment with an anticoagulant;
10. Head injury or open wound that contraindicates use of the Chordate Headband;
11. Known allergy to polyvinylchloride, a material used in the Chordate Catheter, or medicinal liquid paraffin;
12. Concurrent condition or risk of non-compliance that, in the investigator's opinion, may affect the interpretation of performance or safety data or which otherwise contraindicates participation in a clinical investigation;
13. Pregnant and lactating women;
14. Participation in a clinical investigation within 3 months of enrolment or planned participation at any time during this clinical investigation;
15. Previous participation in this study;
16. Employees of the study site or the sponsor directly involved with the conduct of the study, or immediate family members of any such individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arne May, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (10):
- Finland (4):
  - Terveystalo Ruoholahti, Helsinki
  - Helsingin päänsärkykeskus / Aava Itäkeskus, Helsinki
  - Terveystalo Tampere, Tampere
  - Suomen Terveystalo Turku, Turku
- Germany (6):
  - Lewis Neurologie, Stuttgart, Baden-Wurttemberg
  - Neurologie- & Kopfschmerzzentrum, München, Bavaria
  - Klinikum Großhadern / Neurologische Klinik der Universität München, München, Bavaria
  - Migräne-Klinik Königstein, Königstein im Taunus, Hesse
  - Universitätsmedizin Rostock / Klinik und Poliklinik für Neurologie, Rostock, Mecklenburg-Vorpommern
  - CTC North am Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No
Due to uncertainties in EU data protection legislation individual deidentified participant data are not shared. The main uncertainty is the concept of what "deidentified" means. It appears not to mean that the data set of a person is simply separated from the person's name. What additional operations have to be done appears to depend on technological capabilities to re-identify the persons associated with the data set. A common perception is that the technological capabilities for re-identification are permanently increasing. This could have the effect that public data sets that are regarded as deidentified now might become re-identifiable data sets in the future. Once this happens, the sponsor is no longer able to make the publication of the data sets un-happen. This could result in punishment by EU data protection authorities. The sponsor wants to avoid this.

REFERENCES:
- [Derived] Hoffmann J, Kaube H, Rimmele F, Jurgens TP, Nissila M, Gaul C, Kallela M, Keski-Santti P, Sumelahti ML, Straube A, Lewis D, Hoffmann V, Wirtz L, Rempel A, Bohm O, May A. Kinetic Oscillation Stimulation for the Preventive Treatment of Chronic Migraine: A Randomized, Double-Blind, Sham-Controlled Trial. Neurology. 2025 Feb 11;104(3):e210220. doi: 10.1212/WNL.0000000000210220. Epub 2025 Jan 9. PMID 39787477

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment | Sham Treatment
Started | 75 | 69
Randomization | 75 | 69
Safety Analysis Set (SAF) | 76 | 68
Full Analysis Set (FAS) | 71 | 69
Completed | 67 | 65
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Population: One subject was randomized to and treated with placebo and was assigned to the placebo group in the FAS, but received active treatment for a short time at Visit 1 and was therefore assigned to the active group in the SAF. Baseline subject demographics are based on the SAF.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Sham Treatment | Total
Number analyzed (Participants) | 76 | 68 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 67 | 143
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 48 [20 to 64] | 46 [19 to 67] | 48 [19 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 57 | 122
  Male | 11 | 11 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 75 | 68 | 143
  Arabian (Jordan) | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Finland | 25 | 22 | 47
  Germany | 51 | 46 | 97
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (5.6) | 25.3 (5.0) | 25.9 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (4-week Screening Period) in Monthly Headache Days With Moderate to Severe Intensity in 4-week Performance Assessment Period.
Description: Least square mean change from Baseline (4-week screening period) in monthly headache days with moderate to severe intensity in 4-week performance assessment period.
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 14 to Day 42
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: change in days
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 67 | 65
change in days | -3.45 (0.62) | -1.22 (0.62)
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0132, ANCOVA — analysis of covariance (ANCOVA) model containing terms for treatment, baseline value and medication overuse. Group-sequential analysis using updated boundaries from interim analysis; Mean Difference (Final Values) = -2.23, 95% CI 2-sided [-4.11 to -0.49]

2. Secondary Outcome: Mean Change From Baseline in Monthly Headache Days With Moderate to Severe Intensity in Follow-up Period
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 43 to Day 70
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: change in days
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 66 | 65
change in days | -3.15 (0.59) | -0.47 (0.59)
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0014, ANCOVA; ANCOVA model containing terms for treatment, baseline value and medication overuse; Mean Difference (Final Values) = -2.68, 95% CI 2-sided [-4.32 to -1.04]

3. Secondary Outcome: Mean Change From Baseline to Performance Assessment Period in Monthly Migraine Days
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 14 to Day 42
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: change in days
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 67 | 65
change in days | -3.57 (0.60) | -1.17 (0.60)
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0048, ANCOVA; ANCOVA model containing terms for treatment, baseline value and medication overuse; Mean Difference (Final Values) = -2.40, 95% CI 2-sided [-4.06 to -0.73]

4. Secondary Outcome: Mean Change From Baseline to Follow-up Period in Monthly Migraine Days
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 43 to Day 70
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: change in days
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 66 | 65
change in days | -3.72 (0.60) | -0.85 (0.60)
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0008, ANCOVA; ANCOVA model containing terms for treatment, baseline value and medication overuse; Mean Difference (Final Values) = -2.87, 95% CI 2-sided [-4.54 to -1.20]

5. Secondary Outcome: Mean Change From Baseline to Performance Assessment Period in 4-week Headache Days (Mild, Moderate and Severe Intensity) - All Intensities
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 14 to Day 42
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: change in days
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 67 | 65
change in days | -2.88 (0.57) | -1.35 (0.58)
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0598, ANCOVA; ANCOVA model containing terms for treatment, baseline value and medication overuse; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-3.12 to 0.06]

6. Secondary Outcome: Mean Change From Baseline to Follow-up Period in 4-week Headache Days (Mild, Moderate and Severe Intensity) - All Intensities
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 43 to Day 70
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: change in days
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 66 | 65
change in days | -3.65 (0.62) | -1.75 (0.62)
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0310, ANCOVA; ANCOVA model containing terms for treatment, baseline value and medication overuse; Mean Difference (Final Values) = -1.90, 95% CI 2-sided [-3.63 to -0.17]

7. Secondary Outcome: Proportion of Subjects With 30% or Greater Reduction in Headache Days of Moderate to Severe Intensity in Performance Assessment Period
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 14 to Day 42
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 68 | 67
Participants | 32 | 17
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0102, Chi-squared

8. Secondary Outcome: Proportion of Subjects With 30% or Greater Reduction in Headache Days of Moderate to Severe Intensity in Follow-up Period
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 43 to Day 70
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 69 | 67
Participants | 27 | 19
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.1615, Chi-squared

9. Secondary Outcome: Proportion of Subjects With 50% or Greater Reduction of Headache Days of Moderate to Severe Intensity in Performance Assessment Period
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 14 to Day 42
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 68 | 67
Participants | 20 | 11
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0798, Chi-squared

10. Secondary Outcome: Proportion of Subjects With 50% or Greater Reduction of Headache Days of Moderate to Severe Intensity in Follow-up Period
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 43 to Day 70
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 69 | 67
Participants | 16 | 9
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.1300, Chi-squared

11. Secondary Outcome: Change in the Use of Abortive Medication in Performance Assessment Period
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 14 to Day 42
Population: FAS
Measure: Mean (Standard Deviation); unit: change in days
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 67 | 65
change in days | -2.016 (4.565) | -0.857 (4.721)
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0660, Van-Elteren — posthoc; Median Difference (Final Values) = -1.0

12. Secondary Outcome: Change in the Use of Abortive Medication in Follow-up Period
Time Frame: Interval from Day -28 to Day 0 and Interval from Day 43 to Day 70
Population: FAS
Measure: Mean (Standard Deviation); unit: change in days
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 66 | 65
change in days | -2.490 (4.260) | -0.660 (5.552)
Statistical Analysis 1: Comparison: Active Treatment vs Sham Treatment; Test type: Superiority; p = 0.0152, Van-Elteren — posthoc; Median Difference (Final Values) = -2.0

13. Secondary Outcome: Headache Impact Test
Description: The headache impact test-6 (HIT-6) is a 6-item self-administered questionnaire that evaluates the extent of disability a subject experiences due to headache by measuring the subject's level of pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The final total score is obtained from simple summation of the 6 items. The total score ranges between 36 and 78, with larger scores reflecting greater impact.
  Reported is the change from Baseline in the final total score at the respective visit.
Time Frame: Days -28, 0, 14 (Visit 3), 42 (Visit 7), 70 (follow-up)
Population: assessments of individual subjects missing at some visits
Measure: Mean (Standard Deviation); unit: change in score on a scale from Baseline
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 71 | 69
change in score on a scale from Baseline
  Visit 3: number analyzed (Participants) | 69 | 68
  Visit 3 | -2.6 (5.2) | -1.5 (3.1)
  Visit 7: number analyzed (Participants) | 68 | 66
  Visit 7 | -4.1 (6.8) | -2.2 (4.8)
  Follow-up visit: number analyzed (Participants) | 69 | 67
  Follow-up visit | -3.8 (7.4) | -1.7 (5.4)

14. Secondary Outcome: Migraine-Specific Quality of Life Questionnaire (MSQ) - Role Function - Restrictive
Description: The role function-restrictive dimension of the MSQ assesses how migraines limit daily activities and interactions during the past 4 weeks. It includes 7 items. Each item is scored on a 6-point scale ranging from 1 (none of the time) to 6 (all of the time). The scores of these items are summed and then transformed to a 0-100 scale. This means the minimum score of the role function restrictive dimension is 0 and the maximum score is 100 where a higher score indicates a better health status.
  Reported is the change from Baseline in the role function restrictive dimension of the MSQ at the respective visit.
Time Frame: Days -28, 0, 14 (Visit 3), 42 (Visit 7), 70 (follow-up)
Population: assessments of individual subjects missing at some visits
Measure: Mean (Standard Deviation); unit: change in score on a scale from Baseline
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 71 | 69
change in score on a scale from Baseline
  Visit 3: number analyzed (Participants) | 69 | 68
  Visit 3 | 7.4 (16.3) | 5.4 (11.2)
  Visit 7: number analyzed (Participants) | 68 | 66
  Visit 7 | 13.3 (19.9) | 7.5 (17.0)
  Follow-up: number analyzed (Participants) | 68 | 67
  Follow-up | 11.9 (21.4) | 4.9 (19.8)

15. Secondary Outcome: MSQ - Role Function - Preventive
Description: The role function-preventive dimension of the MSQ assesses how migraines prevent from engaging in daily activities during the past 4 weeks. It includes 4 items. Each item is scored on a 6-point scale ranging from 1 (none of the time) to 6 (all of the time). The scores of these items are summed and then transformed to a 0-100 scale. This means the minimum score of the role function-preventive dimension is 0 and the maximum score is 100 where a higher score indicates a better health status.
  Reported is the change from Baseline in the role function-preventive dimension of the MSQ at the respective visit.
Time Frame: Days -28, 0, 14 (Visit 3), 42 (Visit 7), 70 (follow-up)
Population: assessments of individual subjects missing at some visits
Measure: Mean (Standard Deviation); unit: change in score on a scale from Baseline
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 71 | 69
change in score on a scale from Baseline
  Visit 3: number analyzed (Participants) | 69 | 68
  Visit 3 | 4.2 (17.4) | 0.7 (10.9)
  Visit 7: number analyzed (Participants) | 68 | 66
  Visit 7 | 9.2 (20.8) | 4.8 (16.6)
  Follow-up: number analyzed (Participants) | 68 | 67
  Follow-up | 9.8 (22.2) | -0.7 (19.8)

16. Secondary Outcome: MSQ - Emotional Function
Description: The emotional function dimension of the MSQ assesses the emotional impact of migraines during the past 4 weeks. It includes 3 items. Each item is scored on a 6-point scale ranging from 1 (none of the time) to 6 (all of the time). The scores of these items are summed and then transformed to a 0-100 scale. This means the minimum score of the emotional function dimension is 0 and the maximum score is 100 where a higher score indicates a better health status.
  Reported is the change from Baseline in the emotional function dimension of the MSQ at the respective visit.
Time Frame: Days -28, 0, 14 (Visit 3), 42 (Visit 7), 70 (follow-up)
Population: assessments of individual subjects missing at some visits
Measure: Mean (Standard Deviation); unit: change in score on a scale from Baseline
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 71 | 69
change in score on a scale from Baseline
  Visit 3: number analyzed (Participants) | 69 | 68
  Visit 3 | 7.0 (16.2) | 3.0 (14.2)
  Visit 7: number analyzed (Participants) | 68 | 66
  Visit 7 | 10.2 (23.5) | 5.8 (19.2)
  Follow-up: number analyzed (Participants) | 68 | 67
  Follow-up | 11.5 (25.2) | 2.5 (24.7)

17. Secondary Outcome: Patient Global Impression of Severity (PGI-S)
Description: The PGI-S is a 1-item questionnaire to assess the subject's impression of disease severity. The subjects rated the severity of their condition on a scale from 1 to 4: 1=normal, 2=mild, 3=moderate, 4=severe
Time Frame: Days -28 (screening), 0 (visit 1), 14 (Visit 3), 42 (Visit 7), 70 (Follow-up)
Population: assessments of individual subjects missing at some visits
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 71 | 69
Participants
  Screening: Not done | 1 | 0
  Screening: normal | 13 | 13
  Screening: mild | 7 | 4
  Screening: moderate | 25 | 24
  Screening: severe | 25 | 28
  Visit 1: Not done | 2 | 1
  Visit 1: normal | 21 | 20
  Visit 1: mild | 5 | 6
  Visit 1: moderate | 22 | 19
  Visit 1: severe | 21 | 23
  Visit 3: number analyzed (Participants) | 69 | 68
  Visit 3: Not done | 1 | 1
  Visit 3: normal | 22 | 24
  Visit 3: mild | 13 | 9
  Visit 3: moderate | 21 | 20
  Visit 3: severe | 12 | 14
  Visit 7: number analyzed (Participants) | 68 | 67
  Visit 7: Not done | 1 | 1
  Visit 7: normal | 23 | 25
  Visit 7: mild | 17 | 10
  Visit 7: moderate | 21 | 18
  Visit 7: severe | 6 | 13
  Follow-up: number analyzed (Participants) | 69 | 67
  Follow-up: Not done | 0 | 0
  Follow-up: normal | 22 | 23
  Follow-up: mild | 17 | 9
  Follow-up: moderate | 20 | 18
  Follow-up: severe | 10 | 17

18. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: n (%) of patients
Time Frame: Days 0, 7, 14, 21, 28, 35, 42, 70
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 76 | 68
Participants
  Any adverse event | 49 | 41
  Any treatment emergent adverse event | 48 | 41
  any serious treatment emergent adverse event | 1 | 0
  Any treatment emergent adverse event related to medical device | 2 | 5
  Any treatment emergent adverse event related to procedure | 17 | 13

ADVERSE EVENTS:
Time Frame: From Day 0 (during and after the first treatment with the investigational medicinal device) to Day 70 (final follow-up visit), i.e, about 10 weeks
Description: [shortened] The definition of AE in this study does not include adverse experiences observed by the patient or in the patient before the investigational medical device application.
  It does not include anticipated device effects of mild character. It does also not include migraine-associated symptoms.
  All AEs were assessed in terms of seriousness (yes, no), severity, outcome, relationship to the investigational medical device, and relationship to study procedures.
Arm/Group | Active Treatment | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/68
Serious Adverse Events (participants affected / at risk) | 1/76 | 0/68
Other Adverse Events (participants affected / at risk) | 49/76 | 41/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=76) | Sham Treatment (N=68)
foot fracture (Injury, poisoning and procedural complications) | 1 (1) | NA — right metatarsal shaft fracture
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=76) | Sham Treatment (N=68)
Tinnitus (Ear and labyrinth disorders) | 2 (5) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Lacrimation increased (Eye disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0
Diarrhea (Gastrointestinal disorders) | 1 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0
Fatigue (General disorders) | 2 (3) | 0
Corona Virus infection (Infections and infestations) | 4 (4) | 4 (4)
Influenza (Infections and infestations) | 0 | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (6) | 6 (6)
Otitis media (Infections and infestations) | 2 (2) | 0
Root canal infection (Infections and infestations) | 0 | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (5)
Dizziness (Nervous system disorders) | 7 (9) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Epixtaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (10) | 3 (8)
Hypertension (Vascular disorders) | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03400059/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT03400059/SAP_001.pdf